CLINICAL TRIAL: NCT02977013
Title: Anti-Xa Assay Correlation to the Efficacy and Safety of Enoxaparin in the Treatment of Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: Mohamed Sayed Mohamed Abbas (Other)
Responsible Party: Sponsor-Investigator, Mohamed Sayed Mohamed Abbas, Doctor, Al Mouwasat Hospital
Organization: Al Mouwasat Hospital (Other)
Other Study IDs: MSAT-5
Record Dates: First submitted 2016-11-27; First posted 2016-11-30 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Anti-Xa Assay in Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with pulmonary embolism treated with enoxaparin: Anti-Xa assay correlation to the efficacy and safety of enoxaparin in the treatment of pulmonary embolism
  Interventions: Diagnostic Test: Anti-Xa assay

INTERVENTIONS:
Diagnostic Test: Anti-Xa assay — Correlation between anti-Xa assay and the efficacy and safety of enoxaparin in the treatment of pulmonary embolism

SUMMARY:
The aim of the present study is to monitor anticoagulant therapy by anti-Xa assay and correlate its level to the efficacy and safety of enoxaparin in the treatment of pulmonary embolism.

DETAILED DESCRIPTION:
This prospective randomized trial was conducted on 42 patients 18 years of age or older in ICU diagnosed to have pulmonary embolism and confirmed by the presence of intraluminal filling defect in CT pulmonary angiography and treated with subcutaneous enoxaparin 1 mg/kg/12 hours. The study was conducted from August 2013 to September 2016.

All the patients were examined daily over a period of 4 weeks for symptoms and signs of recurrent pulmonary embolism (recurrent pulmonary embolism was diagnosed if the repeat CT angiography revealed a new sudden arterial branch cutoff or a new intraluminal filling defect that was not present on the first angiogram), Platelet count (patients with platelet count less than 50,000/mm3 or those with bleeding and platelet count between 50,000 and 100,000/mm3 are considered having severe thrombocytopenia), bleeding (defined as major overt bleeding requiring blood transfusion > 2 units or marked hemoglobin drop > 2 gm/dl or if the bleeding was intracranial or retroperitoneal) and death (defined as all deaths occurring within the 4 weeks of the study) , Then the results were correlated to anti-Xa assay.

ELIGIBILITY:
Inclusion Criteria:

* Patients in ICU and diagnosed to have pulmonary embolism and confirmed by the presence of intraluminal filling defect in CT pulmonary angiography and treated with subcutaneous enoxaparin 1 mg/kg/12 hours.

Exclusion Criteria:

* Patients who underwent thrombolysis, embolectomy or if they are unfit for anticoagulant therapy because of major bleeding or thrombocytopenia (a platelet count below 100,000 per cubic millimeter). Patients were also excluded if they had impaired kidney function with a serum creatinine level above 2 mg/dl or uncontrolled hypertension (blood pressure > 160/100 mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted on 42 patients in ICU diagnosed to have pulmonary embolism by CT pulmonary angiography and treated by subcutaneous enoxaparin 1 mg/kg every 12 hours. Anticoagulant therapy was followed by anti-Xa assay done 4 hours after the third dose of subcutaneous enoxaparin and the results were correlated to the clinical outcome of the patients as regards complications (recurrent pulmonary embolism, bleeding, low platelet count and death).
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Recurrent pulmonary embolism | 4 Weeks
  Recurrent pulmonary embolism was diagnosed if the repeat CT angiography revealed a new sudden arterial branch cutoff or a new intraluminal filling defect that was not present on the first angiogram.
Platelet count | 4 Weeks
  Patients with platelet count less than 50,000/mm3 or those with bleeding and platelet count between 50,000 and 100,000/mm3 are considered having severe thrombocytopenia
Bleeding | 4 Weeks
  Defined as major overt bleeding requiring blood transfusion > 2 units or marked hemoglobin drop > 2 gm/dl or if the bleeding was intracranial or retroperitoneal
Death | 4 Weeks
  Defined as all deaths occurring within the 4 weeks of the study

REFERENCES:
- [Background] Montalescot G, Collet JP, Tanguy ML, Ankri A, Payot L, Dumaine R, Choussat R, Beygui F, Gallois V, Thomas D. Anti-Xa activity relates to survival and efficacy in unselected acute coronary syndrome patients treated with enoxaparin. Circulation. 2004 Jul 27;110(4):392-8. doi: 10.1161/01.CIR.0000136830.65073.C7. Epub 2004 Jul 12. PMID 15249498